CLINICAL TRIAL: NCT05820230
Title: Changes in the Blood-brain Barrier During Maintenance ECT in Formerly Depressed Patients
Acronym: 3BECT
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Poul Videbech, Professor Poul Videbech, University of Copenhagen
Other Study IDs: H-22039168
Record Dates: First submitted 2023-03-24; First posted 2023-04-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to analyse S100-B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine the effect of electroconvulsive therapy (ECT) on the blood-brain barrier (BBB) in patients who had suffered from depression. We will study the BBB with dynamic contrast enhanced (DCE) MRI before and after treatment with a single ECT in patients currently undergoing ECT. The study is an observational (naturalistic) longitudinal study.

DETAILED DESCRIPTION:
Primary hypothesis

1. The BBB permeability to Gadovist (measured as Ki) temporarily increases in the right and left hippocampus (HC) after a single ECT.

   Secondary hypothesises
2. The volume of the right and left HC increases after a single ECT and the volume increase is positively correlated with the BBB permeability
3. A larger post-ECT increase in systolic blood pressure correlates with a larger increase in BBB permeability in the right and left HC.
4. A larger increase in serum S100-B compared to baseline values is correlated with increased BBB permeability in the right and left HC.

ELIGIBILITY:
Inclusion Criteria:

- We will include patients (age 18-75) currently treated with a series of ECT or maintenance ECT referred to the treatment due to moderate to severe depression according to ICD-10.

Exclusion Criteria:

1. Schizophrenia
2. Psychotic symptoms
3. Any substance use (other than cigarette smoking and alcohol consumption within the recommendations of the Danish National Health Authority) within the last 3 months
4. Risk of suicide making transport or participation in the study hazardous
5. Claustrophobia or severe restlessness
6. Contraindications to DCE-MRI (e.g., metallic implants, increased body temperature, reduced kidney function (estimated Global Filtration Rate (eGFR) of <40 ml/min/1.73 m2), pregnancy)
7. Somatic illness potentially confounding results (e.g., any central nervous system diseases or cancers)
8. Lack of consent to being informed of potential medically important findings on MRI or blood tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a series of ECT or maintenance ECT in a hospital at the Mental health services in the Capital Region of Denmark
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Permeability | Permeability is measured before a single ECT and 0-8 hours after a single ECT
  Change in permeability measured as Ki in the units of ml/100g/min in the right and left hippocampus

CONTACTS AND LOCATIONS:
Overall Officials: Poul Videbech, Professor, Principal Investigator — University of Copenhagen & Mental Health Centre Glostrup
Locations (1):
- Mental Health Services of the Capital Region of Denmaark, Copenhagen, Denmark